CLINICAL TRIAL: NCT03717792
Title: Vascular Liver Disease Evaluation, Follow Up and Non-Invasive Diagnostics Program
Acronym: VALID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, Principal Investigator, University Hospital, Bonn
Other Study IDs: VALID
Record Dates: First submitted 2018-10-20; First posted 2018-10-24 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Vascular Disorder of Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Background Vascular liver disorders (VALDI) are rare diseases, for which knowledge on risk factors, appropriate methods of diagnosis, effect of therapy and prognosis still need to be improved.

Aim of the study This project aims to study risk factors, methods of detection, therapy and prognosis in order to elaborate and disseminate updated recommendations for the optimal management of patients with VALDI.

Design of the study Data on patients will be collected from baseline (the date of diagnosis) up to 3 years. During this period, data on clinical condition, laboratory results, diagnostic tests, interventions and outcome will be collected anonymously using standardised review of medical charts by one special trained investigator. Only patients with VALDI are eligible to participate.

DETAILED DESCRIPTION:
Background Vascular liver disorders (VALDI), including Budd-Chiari syndrome (BCS), non-cirrhotic vascular liver disorders (VLD) and idiopathic non-cirrhotic portal hypertension (INCPH) are rare diseases that mainly affect children and young adults. These diseases are related to alterations in hepatic macrocirculation (hepatic veins, portal vein) or microcirculation (small portal veins, sinusoids or both) in the absence of cirrhosis. Even though various types of VALDI differ in presentation and etiology, they still share in part underlying causes and mechanisms.

Most studies on VALDI aim at clarifying etiology, natural history and management have been retrospective and are based on a relatively small number of patients. A European Union FP5 funded project from 2003 to 2005 (EN-Vie) performed several prospective observational studies, in which 157 patients with BCS and 102 patients with acute VLD were included. However, chronic VLD and INCPH were not included in the EN-Vie project.

Prothrombotic disorders are found in 65 to 85% of patients with BCS or VLD, but only 20-40% of INCPH patients. By contrast, chronic inflammatory conditions are more frequently encountered in patients with INCPH and VLD than in those with BCS. There is evidence for a significant genetic influence in patients with INCPH. Still, in over 40% of INCPH patients the cause remains unknown. The reason for these differences in causes among the various VALDI, as well as the mechanisms for specific sites of thrombosis according to the underlying conditions remain obscure.

VALDI complications mostly consist in gastrointestinal bleeding, refractory ascites, bacterial infections, hepatocellular carcinoma, and ultimately liver failure. Such complications are observed in approximately 60%, 20% and 15% of patients with BCS, VLD and INCPH, respectively. The incidence of bleeding related to portal hypertension is as high as 20 % patients-year in patients with VLD or INCPH. Recurrent or extensive thrombosis may jeopardize liver transplantation or lead to high morbidity and mortality complications, e.g. intestinal infarction. Moreover, complications related to the underlying disorders superimpose on those directly related to VALDI, and particularly so for acquired blood diseases.

The outcome of VALDI has been recently evaluated in large prospective European studies. (a) A recent update on BCS cohort showed a good outcome with a strategy comprising anticoagulation therapy and, when needed, angioplasty, stenting, TIPS, or liver transplantation. Similarly, anticoagulation at the early stage of VLD has been shown to prevent thrombus extension and, in 40% of the cases, to be accompanied by recanalization. The results of these studies have had an impact much beyond the field of primary VALDI. Actually it proved instrumental in developing novel and promising strategies with anticoagulation for the management of cirrhosis, a chronic parenchymal liver disease much more common than VALDI. (b) By contrast, for patients with chronic VLD prospective follow-up data are not available. Retrospective data suggest that anticoagulation is not associated with excessive bleeding. However, in patients at risk for gastrointestinal bleeding due to portal hypertension and a mild or moderate risk of recurrent thrombosis, the benefit-risk ratio of anticoagulation therapy is particularly unclear. Furthermore, the time point, if any, when anticoagulation shifts from a beneficial to a detrimental effect, has not been explored. (c) The natural history of INCPH evaluated in only 3 retrospective surveys indicates that the incidence of extrahepatic VLD is surprisingly high, whereas advanced liver disease or hepatopulmonary syndrome may occur in up to 15% of patients. Therefore, anticoagulation therapy, TIPS and liver transplantation have also been proposed in patients with INCPH.

• Although recent studies have provided a marked impetus to the field of clinical research on VALDI, crucial information is still lacking, particularly in the areas of etiology, inherited factors, and treatment. Etiology is still unknown in 40% of the patients; genetic data are incomplete, therapeutic trials, although badly needed have never been performed, so that recommendations for treatments (with potentially fatal side effects in these high bleeding risk population) rely on limited data.

Aims Identification of incident and prevalent cases of VALDI as a basis for the implementation of future studies, namely interventional randomised control studies, observational studies, and prognostic studies including the identification of new biomarkers for these diseases through the analysis of the prospectively recorded data according to consensual management.

This study will allow to obtain:

Incidence estimates Increased numbers of patients candidates to future studies Homogeneous, robust and consistent criteria for diagnosis, follow-up and treatment, allowing clearly defined cohorts of patients to be constituted.

Identify the collections of biological and tissue samples stored in the same conditions, for future the identification of novel biomarkers. Samples will have to be linked to high quality clinical, laboratory and imaging data for translational studies

Create a basis for continuous collections for a large variety of research purposes including:

Prognostic research Systems biology research including (epi)genetic research Clinical trials using various design adapted for rare diseases Health care policies and cost-effectiveness studies

ELIGIBILITY:
Inclusion Criteria:

* all patients with vascular liver disease

Exclusion Criteria:

* patients without vascular liver disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include all patients above 18 years of age with vascular liver disease diagnosed according to EASL Clinical Practice Guideline.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications of Portal Hypertension | up to 3 years
  Ascites, Varices, Bleeding, Encephalpathy, Thrombosis

SECONDARY OUTCOMES:
Mortality | up to 3 years
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University of Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany